CLINICAL TRIAL: NCT03171051
Title: Feasibility Study of a 950 nm Wavelength LED Device for Non-Invasive Lipolysis of the Flanks
Brief Title: LED Device for Non-Invasive Lipolysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: device development placed on hold
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CS0117
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Lipolysis
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: All subjects to receive the same treatments - right flank of abdomen with the experimental LED device and the left flank of the abdomen with the active comparator diode laser device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Lipolysis treatment (Other): The right flank of the abdomen will be treated with the 950nm LED device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  The left flank of the abdomen will be treated with the 1050nm diode laser device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  Interventions: Device: 950 nm LED Device; Device: 1050nm Diode Laser Device

INTERVENTIONS:
Device: 950 nm LED Device — Device to be used in aesthetic and cosmetic procedures which consists of a console and an applicator belt that delivers the treatment LED to the subject's skin.
Device: 1050nm Diode Laser Device — FDA approved laser device that has been shown to reduce fat in the flanks by heating the fat cells and causing them to burst. The contents of the cells are then cleared naturally by the body.
  Other Names: SculpSure

SUMMARY:
This study is being conducted to evaluate the ability of a light emitting diode (LED) study device's ability to raise the temperatures on flank tissue to a similar level compared to an approved laser device (SculpSure by Cynosure). Laser treatments have been shown to reduce fat in the flanks by heating the fat cells and causing them to burst. The contents of the cells are then cleared naturally by the body.

DETAILED DESCRIPTION:
This is an open-label, feasibility study comparing the tissue temperature profile of a 950 nm LED device and a 1060 nm diode laser for non-invasive lipolysis of the flanks. The study will enroll up to 10 subjects requesting non-invasive lipolysis of the flanks. Each subject will receive a single treatment with each device on opposite flanks. Tissue temperatures in the treated areas will be recorded at various tissue depths and compared. Subjects will be asked to assess their discomfort and pain of the study treatment using a 10 cm visual analog scale (VAS). In addition, the safety (number of treatment related adverse events) of the LED device will be compared to the reference device at the time of treatment and one week later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, male or female, ≥ 18 years of age or older with skin types 1-VI.
* Having moderate excess bilateral fatty tissue of the flanks, suitable area for non-invasive lipolysis.
* Women of child-bearing potential (women who have not had a hysterectomy, bilateral oophorectomy or are not postmenopausal) are required to be using a reliable method of birth control for at least three months prior to enrolment and throughout the course of the study and have a negative urine pregnancy test at baseline.

Exclusion Criteria:

* Pregnant, expectation of pregnancy, postpartum or nursing (<6 months).
* History of skin disease in the area to be treated over the last 6 months.
* Previous surgical intervention to the treatment area.
* History of skin cancer or pre-cancerous lesions at the treatment areas.
* Having any electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* History of immunosuppressive diseases, including AIDS and HIV infection, or use of immunosuppressive medications;
* Uncontrolled systemic diseases such as diabetes.
* Active infections in the treatment area.
* History of dysplastic nevi.
* Significant concurrent skin conditions or any inflammatory skin conditions.
* Active herpes simplex infections (e.g. cold sores), open lacerations or abrasions in the treatment area.
* Chronic or cutaneous viral, fungal, or bacterial diseases.
* Use of Accutane™ (Isotretinoin) within the past six months.
* Keloid or hypertrophic scar formation in the treatment area.
* Tattoos in the treatment area.
* History of auto-immune disorders.
* Erythema abigne, when identified treatments should be discontinued.
* History of photosensitivity disorder that can be exacerbated by laser or intense light.
* Use of medications, herbal supplements, perfumes or cosmetics that may affect sensitivity to light.
* History of poor wound healing in the treatment area.
* Sunburns.
* Unable or unlikely to refrain from artificial tanning, including the use of tanning booths, prior (at least a month) and during the course of the evaluation.
* Prior skin treatment with laser or other devices on the same treatment area within the last six months prior to study enrollment or during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Iger, PhD, Study Director — Venus Concept Ltd.
Locations (1):
- Sadick Research Group, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study. Sharing of IPD may occur if the study supports further development of the device.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lipolysis Treatment: The right flank of the abdomen will be treated with the LED device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  950 nm LED Device: Device to be used in aesthetic and cosmetic procedures which consists of a console and an applicator belt that delivers the treatment LED to the subject's skin.
  The left flank of the abdomen will be treated with the diode laser device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  1050nm Diode Laser Device: FDA approved laser device that has been shown to reduce fat in the flanks by heating the fat cells and causing them to burst. The contents of the cells are then cleared naturally by the body.
Period: Overall Study
Arm/Group | Lipolysis Treatment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subject is receving LED treatment on the right abdomen and Laser treatment on the left abdomen.
Units Other Than Participants: abdomen
Groups:
- Lipolysis Treatment: The right flank of the abdomen will be treated with the LED device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes. No baseline temperatures were obtained.
  The left flank of the abdomen will be treated with the diode laser device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes. No baseline temperatures were obtained.
Arm/Group | Lipolysis Treatment
Number analyzed (Participants) | 10
Number analyzed (abdomen) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Temperature Profile Comparison of the LED Device as Compare to the Reference Device (Diode Laser) at Various Tissue Depths
Description: Immediately (within 2 minutes) after treatment of the area, 3 sterile thermocouple needles of different lengths (9.5-14 mm), will be inserted into the center of each applicator footprint. Temperature readings from each thermocouple needle will be recorded.
Time Frame: At time of treatment
Population: Subject had one side of their abdomen treated with the experimental 950nm LED and the other side of their abdomen treated with the 1050nm diode laser. Note that temperature data was not available for 1 participant for the 1050nm laser at the 9.5mm tissue depth.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Lipolysis Treatment
Number analyzed (Participants) | 10
degrees Celsius
  950nm LED Mean Temperature at 14mm | 44.9 (2.3)
  1050nm Laser Temperature at 14mm | 42.5 (2.6)
  950nm LED Mean Temperature at 9.5mm | 43.9 (2.7)
  1050nm Laser Mean Temperature at 9.5mm: number analyzed (Participants) | 9
  1050nm Laser Mean Temperature at 9.5mm | 41.5 (3.8)

2. Secondary Outcome: Visual Analog Scale (VAS)
Description: Subjects reported level of discomfort and pain after treatment with LED and Laser applicators on a 10 cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of 'no pain at all' (value of 0 cm) and 'worst pain imaginable' (value of 10 cm).
Time Frame: Time of treatment
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Treatment Group: Subjects received two lipolysis treatments: the left flank of the abdomen received treatment with the diode laser device and the right flank of the abdomen received treatment with the LED device.
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
score on a scale
  950nm LED VAS | 4.1 [0.4 to 7.6]
  1050nm Laser VAS | 3.48 [0.3 to 7.7]

ADVERSE EVENTS:
Time Frame: The adverse events were collected from 7 June 2017 until 13 July 2017. All reportable events with start dates occurring any time after informed consent is obtained were followed until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation.
Groups:
- Lipolysis Treatment: The right flank of the abdomen will be treated with the 950nm LED device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  The left flank of the abdomen will be treated with the 1050nm diode laser device. The treatment area will be heated initially for 4 minutes at 41W followed by a duty cycle of 25 sec on and 10 sec off time at 29W for 16 minutes. Total treatment time will be 24 minutes.
  950 nm LED Device: Device to be used in aesthetic and cosmetic procedures which consists of a console and an applicator belt that delivers the treatment LED to the subject's skin.
  1050nm Diode Laser Device: FDA approved laser device that has been shown to reduce fat in the flanks by heating the fat cells and causing them to burst. The contents of the cells are then cleared naturally by the body.
Arm/Group | Lipolysis Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipolysis Treatment (N=10)
inflammatory panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) — Panniculitis resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03171051/Prot_SAP_000.pdf